CLINICAL TRIAL: NCT00848120
Title: An Open Label Study to Evaluate the Safety and Reduction in Signs and Symptoms During Treatment With Tocilizumab in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Study to Assess the Effect of Tocilizumab on Signs and Symptoms in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22074
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks for 24 weeks

SUMMARY:
This single arm, open label study will assess the safety and efficacy, with regard to reduction of signs and symptoms,of treatment with tocilizumab in patients with moderate to severe active rheumatoid arthritis. Patients will receive tocilizumab 8 mg/kg IV every 4 weeks for a total of 6 infusions. Patients already receiving methotrexate at entry into the study may continue with their treatment together with tocilizumab.The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients,>=18 years of age;
* rheumatoid arthritis diagnosed >8 weeks and <4 years prior to baseline;
* naive to, or not responding well to, methotrexate;
* swollen joint count >=8 (66 joint count) and tender joint count>=8 (68 joint count) at screening and baseline.

Exclusion Criteria:

* rheumatic autoimmune disease other than rheumatoid arthritis;
* patients with functional class IV rheumatoid arthritis;
* history of, or current, inflammatory joint disease other than rheumatoid arthritis, or other systemic autoimmune disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-12-31 (Actual); Primary Completion 2010-02-13 (Actual); Study Completion 2010-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Philippines (4):
  - Alabang Medical Center, City of Muntinlupa
  - Manila Doctors Hospital; Rheumatology Section, Manila
  - Jose Reyes Memorial Medical Center, Manila
  - Our Lady of Mount Carmel Medical Center, San Fernando City

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 Milligrams Per Kilogram (mg/kg): Participants received tocilizumab 8 mg/kg intravenously (IV) once every 4 weeks for 24 weeks.
Period: Overall Study
Arm/Group | Tocilizumab 8 Milligrams Per Kilogram (mg/kg)
Started | 29
Completed | 28
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received any part of an infusion of study drug.
  Intent to Treat (ITT) Population was used for efficacy analyses. All participants who have received any part of an infusion of study medication were included in this population.
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg IV once every 4 weeks for 24 weeks.
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Percent (%) Improvement (ACR20 Response) at Week 24
Description: ACR20 response: greater than or equal to (≥) 20% improvement in tender or swollen joint counts and 20% improvement in 3 of the following 5 criteria: 1) Physician's global assessment of disease activity, 2) participant assessment of disease activity, 3) Patient Assessment of Pain (visual analog scale [VAS]), 4) participant assessment of functional disability via a Health Assessment Questionnaire (HAQ), and 5) erythrocyte sedimentation rate (ESR) at each visit.
Time Frame: Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
percentage of participants | 86

2. Secondary Outcome: Percentage of Participants Achieving ACR 50% Improvement (ACR50 Response) at Week 24
Description: ACR50 response: ≥50% improvement in tender or swollen joint counts and 50% improvement in 3 of the following 5 criteria: 1) Physician's global assessment of disease activity, 2) participant assessment of disease activity, 3) Patient Assessment of Pain (VAS), 4) participant assessment of functional disability via a HAQ, and 5) ESR at each visit.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
percentage of participants | 66

3. Secondary Outcome: Percentage of Participants Achieving ACR 70% Improvement (ACR70 Response) at Week 24
Description: ACR70 response: ≥70% improvement in tender or swollen joint counts and 70% improvement in 3 of the following 5 criteria: 1) Physician's global assessment of disease activity, 2) participant assessment of disease activity, 3) Patient Assessment of Pain (VAS), 4) participant assessment of functional disability via a HAQ, and 5) ESR at each visit.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
percentage of participants | 48

4. Secondary Outcome: HAQ Disability Index (HAQ-DI) Score at Baseline and Week 24
Description: HAQ-DI is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty 1=with some difficulty 2=with much difficulty 3=unable to do. To calculate HAQ-DI the participant must have a domain score for at least 6 of 8 domains. The HAQ-DI is the sum of the scores, divided by the number of domains that have a score (in range 6-8) for a total possible score minimum/maximum 0 (best) to 3 (worst).
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
units on a scale
  Baseline | 0.75 (0.53)
  Week 24 | 0.23 (0.31)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Week 24 versus baseline; Test type: Superiority or Other; p < 0.001, ANOVA

5. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score at Baseline and Week 24
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participants response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the health status.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
units on a scale
  Baseline | 1.93 (0.61)
  Week 24 | 1.03 (0.46)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Week 24 versus baseline; Test type: Superiority or Other; p < 0.001, ANOVA

6. Secondary Outcome: Disease Activity Score Based on 28 Joint Count - Erythrocyte Sedimentation Rate (DAS28-ESR) at Baseline and Week 24
Description: DAS28-ESR calculated from the number of swollen joints and tender joints using the 28 joints count, the ESR (millimeters per hour [mm/hour]) and Patient's Global Assessment of disease activity (participant rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 less than or equal to (≤)3.2 equals (=) low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
units on a scale
  Baseline | 6.94 (0.53)
  Week 24 | 2.73 (0.93)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Week 24 versus baseline; Test type: Superiority or Other; p = 0.001, ANOVA

7. Secondary Outcome: Percentage of Participants With Disease Remission at Week 24 Assessed Using DAS28-ESR
Description: DAS28-ESR calculated from the number of swollen joints and tender joints using the 28 joints count, the ESR (mm/hour) and Patient's Global Assessment of disease activity (participant rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 <2.6=remission.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
percentage of participants | 34

8. Secondary Outcome: Percentage of Participants With Low Disease Activity at Week 24 Assessed Using DAS28-ESR
Description: DAS28-ESR calculated from the number of swollen joints and tender joints using the 28 joints count, the ESR (mm/hour) and Patient's Global Assessment of disease activity (participant rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 >2.6 and <3.2=low disease activity.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
percentage of participants | 45

9. Secondary Outcome: Time to Onset of ACR20/50/70 Response
Description: Time to onset of ACR 20/50/70 response was calculated as the number of weeks from the administration of the first dose of study drug until the date of first achievement of ACR 20/50/70 per criteria.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 29
weeks
  ACR20 | 4 [4 to 8]
  ACR50 | 12 [8 to 24]
  ACR70 | 24 [16 to NA] — The 3rd quartile range could not be estimated because less than 75% of participants achieved ACR70.

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of screening until 4 weeks after the last infusion.
Arm/Group | Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 24/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab 8 mg/kg (N=29)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=29)
Elevated AST/SGOT level (Metabolism and nutrition disorders) | 24
Elevated ALT/SGPT level (Metabolism and nutrition disorders) | 20
Elevated AST ad ALT levels (Metabolism and nutrition disorders) | 3
Urinary tract infection (UTI) (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Systemic viral infection (Infections and infestations) | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 1
Fatty liver (Hepatobiliary disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colonic diverticulitis (Gastrointestinal disorders) | 1
Internal hemorrhoids, grade 1 (Gastrointestinal disorders) | 1
Non ulcer dyspepsia (Gastrointestinal disorders) | 1
Pruritic back (Skin and subcutaneous tissue disorders) | 1
Pruritic, erythematous scaly plaques over interdigital areas (right foot, first-third toes) (Skin and subcutaneous tissue disorders) | 1
Rashes on chest: back (Skin and subcutaneous tissue disorders) | 1
Rashes on toes (Skin and subcutaneous tissue disorders) | 1
Erythematous, pruritic maculopapular rash (Skin and subcutaneous tissue disorders) | 1
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1
Carpal tunnel syndrome (R) (Nervous system disorders) | 1
Trigger finger 4th digit left hand (Musculoskeletal and connective tissue disorders) | 1
Uterine myoma with nabothian cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Paresthesia at the palm of infusion (Nervous system disorders) | 1
Knee effusion (Musculoskeletal and connective tissue disorders) | 1
Chills and increased pain (General disorders) | 1
Headache/back pain (General disorders) | 1
Fever and headache (General disorders) | 1
Cough productive due to infection (Respiratory, thoracic and mediastinal disorders) | 1
Acute pharyngitis probably viral etiology (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Dengue (Infections and infestations) | 1
Folliculitis left ear (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.